CLINICAL TRIAL: NCT02165085
Title: Identification of Plasmatic Biomarkers in Vascular Ehlers-Danlos Syndrome
Brief Title: Biomarkers in Vascular Ehlers-Danlos Syndrome
Acronym: MEDIC
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P110907
Record Dates: First submitted 2014-05-07; First posted 2014-06-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Vascular Ehlers-Danlos Syndrome
Keywords: Biomarkers; Ehlers-Danlos syndrome, vascular type; Pathophysiology
MeSH Terms: conditions — Ehlers-Danlos Syndrome, Type IV

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, Plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Vascular-Ehlers Danlos syndrome: N=50 patients with vascular Ehlers-Danlos syndrome
- Spontaneous arterial dissection(s): N=50 patients
- Healthy volunteers: n=100 Healthy volunteers

SUMMARY:
The purpose of this study is to determine whether patients with vascular Ehlers-Danlos syndrome present significant and specific changes of arterial endothelial and smooth muscular cell signalling/secretion, in comparison to matched healthy volunteers and patients with spontaneous arterial dissections.

DETAILED DESCRIPTION:
Vascular Ehlers-Danlos syndrome is a rare inherited disease which confers exceptional organ fragility in seamingly healthy young adults. The disease is caused by a mutation in the COL3A1 gene encoding type III collagen, critical to ensure physical resistance to mechanical stress of hollow organs. The disease results in increased tissular fragility, responsible of spontaneous arterial ruptures and dissections and spontaneous bowel perforations. The life-expectancy of patients with vascular Ehlers-Danlos syndrome is reduced by these recurring accidents. The exact mechanisms that trigger arterial accidents are unknown. Recent findings suggest a possible deleterious effect of inflammation and a possible dysregulation of the TGF-beta pathway. Thus, the purpose of this study is to identify further alterations in vascular endothelial and smooth muscular cell signalling/secretion, and to confirm previously suggested mechanisms of arterial accidents in vEDS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with vascular Ehlers-Danlos syndrome must have been positively tested for a pathogenic mutation within the COL3A1 gene.
* In patients with arterial dissection(s) any associated systemic arterial disease must have been ruled out, especially vascular Ehers-Danlos syndrome

Exclusion Criteria:

-All subjects must not present any chronic systemic disease, any acute disease within seven days prior to enrollment, diabetes mellitus and arterial hypertension.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with vascular Ehlers-Danlos syndrome and patients with spontaneous dissection(s) will be recruited from the French National Referral Centre for Rare arterial diseases, Hopital Europeen Georges Pompidou, Paris, France. Healthy volunteers will be recruited by the clinical investigations center, Hopital Europeen Georges Pompidou, Paris, France (random community sample).
Sampling Method: Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2013-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Diagnostic value of plasma biomarkers SEDv | At the end of study (2 years after period of inclusion for first patient)
  Analysis of the diagnostic value of different levels of plasma concentrations of microRNAs

SECONDARY OUTCOMES:
Reference value of biomarkers | At the end of study (2 years after period of inclusion for first patient)
  Compare patients with controls SEDv and two populations (patients with arterial accident spontaneous and healthy volunteers):microRNAs, the expression of circulating markers of tissue remodeling (plasma procollagen type I and III), the expression of a marker of inflammation (sensitivity C-reactive protein CRPus)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Frank, MD, Principal Investigator — Centre de Reference des Maladies Vasculaires Rares, Hopital Europeen Georges Pompidou, APHP, Paris France
Locations (1):
- Hopital europeen Georges Pompidou, Paris, France

REFERENCES:
- [Background] Morissette R, Schoenhoff F, Xu Z, Shilane DA, Griswold BF, Chen W, Yang J, Zhu J, Fert-Bober J, Sloper L, Lehman J, Commins N, Van Eyk JE, McDonnell NB. Transforming growth factor-beta and inflammation in vascular (type IV) Ehlers-Danlos syndrome. Circ Cardiovasc Genet. 2014 Feb;7(1):80-8. doi: 10.1161/CIRCGENETICS.113.000280. Epub 2014 Jan 6. PMID 24399159
- See also: Click here for more information about this disease Vascular Ehlers-Danlos Syndrome — http://www.maladiesvasculairesrares.com